CLINICAL TRIAL: NCT05786352
Title: Outcomes of Enhanced Recovery After Surgery (ERAS) vs. Standard of Care in Cesarean Deliveries: A Randomized-Controlled Trial
Brief Title: Outcomes of Enhanced Recovery After Cesarean (ERAC) Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, gizem boz izceyhan, Gizem Boz İzceyhan, MD, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 141
Record Dates: First submitted 2023-03-04; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Cesarean Section Complications; ERAS
Keywords: ERAS; ERAC

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS (Experimental): ERAS Protocol
  Preoperative:
  1. Clear carbohydrate ( pulp free juice) drink 4 hours before cesarean. Water drinking is allowed until 4 hours before cesarean.
  2. Prophylactic antibiotics 1 hour before cesarean ( Cephazole 2 g iv)
  Intraoperative:
  1. Hypothermia prevention (warming devices)
  2. Pneuomatic compression stockings
  3. Skin preparation with clorhexidine-alcohol
  4. Vaginal preparation with povidone-iodine solution
  Postoperative:
  1. Regular diet within 2 hours after cesarean
  2. Sugar-free gum chewing at postoperative 3rd, 5th and 7th hours, for 20 minutes
  3. Tight control of capillary blood glucose
  4. Mobilization at postoperative 4th hour.
  5. Urinary catheter removal at postoperative 4th hour
  6. Pneuomatic compression stockings
  7. Prevention of nausea and vomiting with routine use of Metoclopramide.
  8. Routine analgesia with Diclofenac sodium suppository application and oral Paracetamole.
  Interventions: Procedure: ERAS protocol
- SOC (Standard of Care) (No Intervention): Preoperative:
  1. Fasting until 6 hours before cesarean.
  2. Prophylactic antibiotics post-delivery during cesarean per institutional protocol ( Cephazole 2 g iv)
  Intraoperative:
  1. Pneuomatic compression stockings as needed
  2. Skin preparation with povidone-iodine solution
  Postoperative:
  1. Water intake at 4th hour after cesarean, traditional delayed feeding until return of intestinal function (bowel sounds or flatus)
  2. Capillary glucose control
  3. Mobilization at postoperative 6th hour.
  4. Urinary catheter removal at postoperative 6th hour
  5. Pneuomatic compression stockings as needed.
  6. Analgesia with Diclofenac sodium intramuscular and oral Paracetamole as needed.

INTERVENTIONS:
Procedure: ERAS protocol — The combination of interventions explained in arm descriptions.
  Arms: ERAS

SUMMARY:
In recent years, a set of evidence-based recommendations called Enhanced Recovery After Surgery (ERAS) is being applied for care of cesarean sections. The effectiveness of ERAS in reducing the length of hospitalization, postoperative complications, the need for analgesics right away after surgery, and the financial cost in the context of cesarean sections has been shown in several studies. There is strong evidence that following ERAS protocols aids postoperative recovery positively. This will be a randomized trial to determine if there is a difference regarding adverse maternal outcomes between ERAS group and standard of care.

DETAILED DESCRIPTION:
Cesarean section is one of the most common surgeries performed today with over one million performed in the United States annually. Our institiution is a tertiary maternity hospital with approximately 3500 cesarean sections annually. A standardized set of guidelines known as Enhanced Recovery After Surgery (ERAS) has been used in a variety of surgical specialties, including colorectal, urologic, gynecologic, and hepatobiliary surgery. The adoption of ERAS guidelines for the obstetric population now offers evidence-based recommendations for postoperative care following cesarean delivery.

At our institution, due to large volume of cesarean section, we encounter a variety of postoperative complications. Institutional standard of care for preoperative, intraoperative and postoperative care has been applied by all providers. In light of recent positive evidence when ERAS protocol is applied, our team aimed to design a randomized controlled trial for comparison of maternal outcomes in ERAS and standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who had cesarean delivery
* Gestational age >37/0 weeks

Exclusion Criteria:

* Diabetes
* Placenta accreta spectrum
* Hypertensive disorders of pregnancy
* Placental abruption
* Need for emergent/urgent cesarean
* Pregnancy complicated by an active infection
* History of allergic reaction to diclofenac sodium, paracetamol or metoclopramide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse composite outcome | Within postoperative 48 hours
  One or more of the following: Prolonged length of hospital stay, infectious complication (urinary tract, wound complications etc.), gastrointestinal complications (need for additional treatment for nausea-vomiting, delayed return of intestinal function, ileus etc.), thrombotic complications, readmission

SECONDARY OUTCOMES:
Postoperative pain | At post operative 6th and 24th hour
  Evaluated with visual analog scale (VAS) A pain scoring scale between 0-10 points, where 0 indicates no pain and 10 indicates the worst pain
Quality of recovery | Immediately before discharge
  Evaluated with Quality of recovery-15 (QoR-15) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women and Children's Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No